CLINICAL TRIAL: NCT04780958
Title: The Effect of Retinol and RBP Levels of Cord Blood and Mothers on Mortality and Morbidity in Prematures With 30 Weeks and Lower
Brief Title: Retinol Status in Preterm Infants and Mothers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Kadir Şerafettin Tekgündüz, Assoc. Prof., Ataturk University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TTU-2020-8630
Record Dates: First submitted 2021-02-24; First posted 2021-03-04 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Vitamin A Deficiency
Keywords: Retinol; Preterm infant; Morbidity; Placenta
MeSH Terms: conditions — Vitamin A Deficiency; Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study population (Other): During the study period, babies born at this hospital with a gestational week of <30 were included .
  Interventions: Other: Serum retinol and RBP levels were determined by enzyme-linked immunosorbent assay.

INTERVENTIONS:
Other: Serum retinol and RBP levels were determined by enzyme-linked immunosorbent assay. — Umbilical cord blood was drawn at birth in all babies included in the study by experienced individuals using a vacutainer. Approximately 6 ml of venous blood was also drawn from the antecubital region of the mothers immediately after the birth in a biochemistry tube.In the serum samples, the retinol levels were analyzed using ELISA kits from the Bioassay Technology Laboratory ( E1548 Hu Jiaxing, Zhejiang, China), RBP levels were analyzed using ELISA kits of Elabscience (E-EL-H1581 Texas USA) following the standard protocol suggested by the manufacturer at the Dynex automated ELISA reading device (Dynex Technologies Headquarters, Chantilly, USA)

SUMMARY:
Retinol and retinol binding protein were studied in the umbilical cord blood of 44 preterm infants with gestation age of < 30 weeks. Serum retinol and RBP levels were determined by enzyme-linked immunosorbent assay. The rate of transplacental retinol passage was calculated. The demographic data of mother and baby, vitamin use in the mother, antenatal steroid application and diseases diagnosed during pregnancy were recorded. An evaluation was made of the retinol, RBP and factors of the mother and baby affecting the transplacental retinol passage. The relationship between retinol and retinol binding protein levels and neonatal mortality and morbidity was investigated.

DETAILED DESCRIPTION:
Study Population Babies born at this hospital with a gestational week of <30 were included in the study. Patients were excluded in the presence of a major abnormality or known congenital metabolic disease in the mother or baby, and the presence of chronic liver, kidney or gastrointestinal system disease in the mother, or if the family did not give consent. A record was made of the gender and birth weight of the babies and gestation week, maternal age, gravidity, status of vitamin intake and use of vitamin A during pregnancy, and antenatal steroid administration in the mothers. A record was made of the presence of early membrane rupture (EMR) diagnosed during the present pregnancy of the mother, preeclampsia/eclampsia, pregnancy-induced hypertension, urinary infection, gestational diabetes mellitus and anemia, if present. We recorded also neonatal mortality and morbidity such as respiratory distress syndrome, retinopathy of prematurity, necrotizing enterocolitis, intraventricular hemorrhage, bronchopulmonary dysplasia,

Sampling and Test Study Method Umbilical cord blood was drawn at birth in all babies included in the study by experienced individuals using a vacutainer. Approximately 6 ml of venous blood was also drawn from the antecubital region of the mothers immediately after the birth in a biochemistry tube, and centrifuged for 10 minutes at 4500 rpm after the completion of coagulation, and the sera were separated. Serum samples were frozen and stored at -80° until the analysis was performed. For the analysis, serum samples were thawed in appropriate circumstances and all analyzes were performed at the Medical Biochemistry Laboratory of Atatürk University at a single session.

In the serum samples, the retinol levels were analyzed using ELISA kits from the Bioassay Technology Laboratory ( E1548 Hu Jiaxing, Zhejiang, China), RBP levels were analyzed using ELISA kits of Elabscience (E-EL-H1581 Texas USA) following the standard protocol suggested by the manufacturer at the Dynex automated ELISA reading device (Dynex Technologies Headquarters, Chantilly, USA). The measurement range of the kit for retinol and RBP was 2ng/ml- 800 ng/ml and 0,07 - 100 ng/mL, respectively.

The formula "umbilical cord retinol/maternal retinol x100" was used for the calculation of placental retinol passage rate in order to show the percentage of maternal retinol passing to the umbilical cord .

Retinol deficiency was evaluated according to the WHO data. A level of < 20 µg/dl was accepted as a deficiency. The level of deficiency was accepted as < 200 ng/ml since the unit used in this present study was ng/ml.

ELIGIBILITY:
Inclusion Criteria:

* Babies born l with a gestational week of <30 and their mothers were included in the study.

Exclusion Criteria:

* Patients were excluded in the presence of a major abnormality or known congenital metabolic disease in the mother or baby, and the presence of chronic liver, kidney or gastrointestinal system disease in the mother, or if the family did not give consent.

Ages: 5 Minutes to 10 Minutes | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Retinol deficiency status in preterm infants and mothers | 4 months
  Number of Participants with retinol deficiency was evaluated according to the WHO data. Concentration of retinol level < 20 µg/dl was accepted as a deficiency. The level of deficiency was accepted as < 200 ng/ml since the unit used in this present study was ng/ml.
Retinol deficiency in preterm infants with respiratory distress syndrome | 3 months
  Numbers of preterm infants with respiratory distress syndrome as assessed accordingly European Consensus Respiratory Distress Syndrome, and have been reported retinol deficiency according to WHO data .
Retinol deficiency in preterm infants with retinopathy of prematurity | 3 months
  Numbers of preterm infants with retinopathy of prematurity as assessed accordingly the International Classification of Retinopathy of Prematurity, and have been reported retinol deficiency according to WHO data .
Retinol deficiency in preterm infants with bronchopulmonary dysplasia | 3 months
  Numbers of preterm infants with bronchopulmonary dysplasia as assessed accordingly the 2001 National Institutes of Health (NIH) Workshop, and have been reported retinol deficiency according to WHO data .
Retinol deficiency in preterm infants with intraventricular hemorrhage | 3 months
  Numbers of preterm infants with intraventricular hemorrhage as assessed accordingly Grading System for Neonatal Intraventricular Hemorrhage, and have been reported retinol deficiency according to WHO data .
Mortality of preterm infants | 3 months
  It was planned to check mortality rate in preterm infants with retinol deficiency. Retinol deficiency rate was calculated accordingly Who data.

CONTACTS AND LOCATIONS:
Overall Officials: Kadir Ş Tekgündüz, Assoc.Prof, Study Director — Ataturk University
Locations (1):
- Ataturk University Medical Faculty, Erzurum, Turkey (Türkiye)